CLINICAL TRIAL: NCT04450199
Title: Does Supplementing Vitamin D Deficiency Affect Fusion Healing Rates in Elective Foot and Ankle Surgery?
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute) (Other)
Collaborators: The Podiatry Foundation (Unknown)
Responsible Party: Principal Investigator, Alan Catanzariti, Program Director, Foot and Ankle Residency Training Program, Allegheny Singer Research Institute (also known as Allegheny Health Network Research Institute)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-126
Record Dates: First submitted 2020-06-11; First posted 2020-06-29 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2023-08

CONDITIONS: Vitamin D Deficiency
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Ergocalciferols; Vitamin D

STUDY DESIGN:
Intervention Model Description: The specific aim of this study is to assess if vitamin D status in the elective foot and ankle fusion population affects fusion healing rates. With this information the investigators hope to ascertain if vitamin D supplementation in the perioperative period leads to superior fusion rates than does no supplementation.
Who Masked: Participant
Masking Description: The patients will be blinded for the duration of the study. This will be accomplished by providing the patients with over encapsulated vitamin D and placebo in pill bottles. Twelve (12) over encapsulated 50,000 IU vitamin D2 or placebo tablets will be packaged in pill bottles for patient use. The Foot & Ankle Institute CRC will document which drug the patients received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Vitamin D (Active Comparator): 12 over encapsulated 50,000 IU Vitamin D2
  Interventions: Drug: Vitamin D2
- Placebo (Placebo Comparator): 12 over encapsulated placebo tablets
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vitamin D2 — Vitamin D tablets
  Other Names: Vitamin D
  Arms: Vitamin D
Other: Placebo — Over encapsulated sugar pills
  Arms: Placebo

SUMMARY:
To assess if vitamin D status in the elective foot and ankle fusion population affects fusion healing categorically (fused vs. un-fused).

DETAILED DESCRIPTION:
This study will be a randomized, 1:1 placebo controlled, blinded, prospective study of level I evidence. The investigators will recruit patients undergoing a major ankle, hindfoot, or midfoot arthrodesis and obtain serum vitamin D levels. Patients that are vitamin D deficient (<30 ng/mL) will then be randomized into two treatment groups: vitamin D supplementation (50,000 IU D2) and no vitamin D supplementation, receiving placebo. Vitamin D levels will be drawn on the day of surgery and 6-8 weeks post-operatively. Outcome variables tested in this study are as follows: bone fusion as an event, time to bone fusion, VAS, and SF-36.

The study will be conducted at 4 investigative sites within the Allegheny Health Network; West Penn Hospital, Forbes Regional Hospital, Twin Towers and Steel Valley Orthopedics & Sports Medicine, Jefferson Hills, PA. Recruitment will stop when approximately 150 subjects are entering the follow-up phase of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females age 18 to 89 years undergoing ankle, hindfoot, or midfoot arthrodesis surgery
2. Vitamin D serum level <30 ng/mL including those concurrently taking vitamin D
3. Ambulatory
4. Women 18 years of age must have a negative urine/serum pregnancy test and must use an acceptable method of contraception, including abstinence, a barrier method (diaphragm or condom), Depo-Provera, or an oral contraceptive, for the duration of the study.

Exclusion Criteria:

1. Revision surgery
2. Tobacco use which has been shown to affect bone healing and increase risk of nonunion
3. Laboratory abnormalities that indicate clinically significant hematologic, hepatobiliary, or renal disease (EXAMPLE below):

   AST/SGOT > 2.0 times the upper limit of normal ALT/SGPT > 2.0 times the upper limit of normal Total bilirubin > 2.0 times the upper limit of normal Hemoglobin < 9 gm/dL White blood cell count < 3,000/ mm3 Platelet count < 100,000/mm3 Creatinine > 2.0 times the upper limit of normal
4. Preexisting disorders known to adversely affect bone healing (e.g. diabetes mellitus with HbA1C greater than or equal to 7, peripheral vascular disease, certain connective tissue disorders, and congenital or acquired disorders of bone metabolism)
5. Preexisting disorders affecting Vitamin D metabolism and/or calcium phosphate homeostasis (e.g. renal failure, hepatic failure, congenital defects in vitamin D metabolism, parathyroid disorders, conditions causing abnormal calcium and/or phosphate absorption)
6. Open wounds to lower extremities which has been shown to increase risk of infection and nonunion
7. Any investigational drug use within 30 days prior to enrollment.
8. Participation in ongoing clinical research
9. Pregnant or lactating females.
10. Patients who are unable to swallow due to acuity of illness or physiologic reason
11. Patients who are unable to provide consent for the study including inability to read or speak English
12. Prisoners who are patients because of their vulnerable population and inability to follow-up
13. Subjects who, in the opinion of the Investigator, may be non-compliant with study schedules or procedures.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-11 (Actual)

PRIMARY OUTCOMES:
Time to Union | 9 months
  Arthrodesis Union using radiographic union determined by independent reviewers

SECONDARY OUTCOMES:
Patient Reported Outcomes SF-36 Questionnaire | 9 months
  Change in patient reported SF-36 questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Patient Reported Outcomes VAS Survey Scores | 9 months
  Change in patient reported VAS survey scores. The scale shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". ... The fifth face represents a pain score of 8, and indicates "hurts a whole lot"; the sixth face represents a pain score of 10, and indicates "hurts worst."

CONTACTS AND LOCATIONS:
Overall Officials: Alan R Catanzariti, DPM, FACFAS, Principal Investigator — The Foot & Ankle Institute, West Penn Hospital
Locations (1):
- The Foot & Ankle Institute/Western Pennsylvania Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
This study has plans for publication and presentation to include a specialized peer reviewed international scientific journal and national conference, respectively. The Principal Investigator and Co-Investigator are part of the AHN and will have complete access to all data for the purpose of publication at study completion. Thanks to the generosity of funding from The Podiatry Foundation of Ohio, making this study possible.